CLINICAL TRIAL: NCT04289857
Title: Efficacy of a Physiotherapy Intervention by Means of Neurodynamic Technique to Improve the Functionality of the Jump in Trampoline Jump Gymnasts. A Randomized Clinical Study.
Brief Title: Neurodynamics to Improve Jump Functionality in Trampoline Jump Gymnasts
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Lockdown
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Neuro
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Athlete Foot
Keywords: Gymnastics trampoline; Neurodynamics; Jump; Range of motion; Randomized clinical trial
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session will last a maximum of 5 minutes, taking place for 3 days a week, over a period of 4 weeks. The intervention will be performed at the start of training (before warm-up).
  Interventions: Other: Neurodynamic training
- Control group (No Intervention): Athletes included in the control group will not perform any intervention, continuing with their usual routine.

INTERVENTIONS:
Other: Neurodynamic training — Starting from a sitting position on a stretcher, with dorsolumbar flexion, it is required to maintain that posture throughout the exercise. Sliding with the straight leg sitting consists of performing alternate movements. First, knee extension and dorsal ankle flexion will be performed, increasing neural tension, combined with cervical extension (to decrease neural tension) in the first instance. Subsequently, knee flexion and plantar ankle flexion (decreasing neural tension) combined with cervical flexion (increasing neural tension) will be performed. The dosage of the technique will be: two seconds for each movement, with 10 repetitions of each one. All sessions will be led by one of the group's researchers.
  Arms: Experimental group

SUMMARY:
The goal of neurodynamics is to restore homeostasis of peripheral nerves. In the current context there is varied evidence that links neurodynamics with clinical pain treatments or different pathologies, but little evidence regarding changes in the functionality of athletes, which could be related to improvements in performance.

The main objective of the study is to determine if the neurodynamic technique is effective in increasing the range of hip mobility and in increasing the jump with counter movement.

Randomized, simple blind clinical study. 15 trampoline jumping gymnasts will be randomized to the two study groups: experimental (active sciatic neurodynamics techniques) and control (without intervention). The intervention will last 4 weeks, with 3 weekly sessions of approximately 5 minutes each. The study variables will be the range of hip flexion movement (goniometry) and the countermove jump (My Jump® application). A descriptive statistical analysis will be performed calculating the main statistical characteristics. The sample distribution will be calculated using a Shapiro-Wills analysis. The changes after each evaluation will be analyzed with the t-student test and with an ANOVA of repeated measures the intra and intersubject effect will be observed. The effect size will be calculated using Cohen's formula.

It is intended to observe improvement in the range of hip flexion movement and in the jump with countermovement.

ELIGIBILITY:
Inclusion Criteria:

* Trampoline jumping gymnasts
* Male
* Aged between 18 and 30 years
* Who train at least 2 days a week
* Federated in the Madrid Gymnastics Federation

Exclusion Criteria:

* Subjects who have a medical diagnosis of musculoskeletal pathology at the time of beginning the study
* Neural pathology in the last 6 months
* With cognitive deficit that prevents them from understanding physical tests and questionnaires
* Have not signed the informed consent

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline hip flexion after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Using a universal goniometer. The subject will be placed supine on a stretcher, identifying the lateral condyle of the femur with a marker, as well as the head of the fibula and the fibular malleolus. The goniometer axis will be placed on the projection of the greater trochanter of the femur. One of the arms of the goniometer arms will be placed parallel to the table (checked with a level). The athlete will be asked for active hip flexion by keeping the knee and ankle in the extended position, being careful not to bend the knee, or swing the pelvis backwards and without turning the hip to external rotation. The other arm of the goniometer will be placed in the direction of the line between the head of the fibula and the fibular malleolus. The unit of measure is the degree, a numerical value whose normal range is 0º-120º

SECONDARY OUTCOMES:
Change from baseline jump height with counter movement after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done with the My Jump application. The athlete will be placed in standing position, with the feet separated at shoulder height and will be asked to jump as high as possible with a rapid movement in countermovement. The hands will remain on the hips during the execution of the jump. The depth of the counter movement will be self-selected and gymnasts will be asked to land near the initial jump zone. They will be instructed verbally to jump as high as possible without specifying the angle of flexion of the knee during the countermovement phase. With the My Jump application, the athlete will be recorded performing the jump with counter movement and the application will determine the height of the jump. The unit of measure is centimeters, where the greater the distance, the greater the height.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain